CLINICAL TRIAL: NCT00974090
Title: A Phase III Study of MP-513 in Combination With Sulfonylurea in Japanese Patients With Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety Study of MP-513 in Combination With Sulfonylurea in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3000-A6
Record Dates: First submitted 2009-09-08; First posted 2009-09-10 (Estimated); Results first posted 2014-05-08 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — 3-(4-(4-(3-methyl-1-phenyl-1H-pyrazol-5-yl)piperazin-1-yl)pyrrolidin-2-ylcarbonyl)thiazolidine; Sulfonylurea Compounds; glimepiride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo / Teneli + SU (Placebo Comparator)
  Interventions: Drug: Placebo / Teneli (Teneligliptin) + SU (Sulfonylurea)
- Teneli / Teneli + SU (Experimental)
  Interventions: Drug: Teneli / Teneli + SU

INTERVENTIONS:
Drug: Placebo / Teneli (Teneligliptin) + SU (Sulfonylurea) — Placebo for 12 weeks (double-blind period) followed by teneligliptin for an additional 40 weeks (open-label period) in combination with sulfonylurea
  Other Names: MP-513; Amaryl; glimepiride
  Arms: Placebo / Teneli + SU
Drug: Teneli / Teneli + SU — Teneligliptin for 12 weeks (double-blind period) followed by teneligliptin for an additional 40 weeks (open-label period) in combination with sulfonylurea
  Other Names: MP-513; Amaryl; glimepiride
  Arms: Teneli / Teneli + SU

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of MP-513 (Teneligliptin) in combination with Sulfonylurea in patients with type 2 Diabetes for 12 weeks administration and to evaluate the safety and efficacy of MP-513 in combination with Sulfonylurea with an extension treatment for up to 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 20 - 75 years old
* Patients who are under dietary management and taking therapeutic exercise for diabetes over 12 weeks before administration of investigational drug
* Patients whose HbA1c is between 7.0% and 10.0%
* Patients who took Sulfonylurea for diabetes over 12 weeks before administration of investigational drug
* Patients who were not administered diabetes therapeutic drugs prohibited for concomitant use within 12 weeks before administration of investigational drug

Exclusion Criteria:

* Patients with type 1 diabetes, diabetes mellitus caused by pancreas impairment, or secondary diabetes (Cushing disease, acromegaly, etc)
* Patients with Class III/IV heart failure symptoms according to NYHA functional classification
* Patients who are gastrointestinal disorder (diarrhea, vomiting)
* Patients with serious diabetic complications
* Patients who are the excessive alcohol addicts
* Patients with severe hepatic disorder or severe renal disorder
* Patients who are pregnant, lactating, and probably pregnant patients, and patients who can not agree to contraception

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2009-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takashi Kadowaki, Professor, Study Director — Tokyo University; Kazuoki Kondo, MD, Study Director — Tanabe Pharma Corporation
Locations (1):
- Sapporo, Hokkaido, Japan

REFERENCES:
- [Background] Kadowaki T, Kondo K. Efficacy and safety of teneligliptin added to glimepiride in Japanese patients with type 2 diabetes mellitus: a randomized, double-blind, placebo-controlled study with an open-label, long-term extension. Diabetes Obes Metab. 2014 May;16(5):418-25. doi: 10.1111/dom.12235. Epub 2013 Dec 10. PMID 24205974

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo / Teneli + SU: Placebo for 12 weeks (double-blind period) followed by teneligliptin for an additional 40 weeks (open-label period) in combination with glimepiride
- Teneli / Teneli + SU: Teneligliptin for 12 weeks (double-blind period) followed by teneligliptin for an additional 40 weeks (open-label period) in combination with glimepiride
Period: Period 1: Double Blind Period
Arm/Group | Placebo / Teneli + SU | Teneli / Teneli + SU
Started | 98 | 96
Completed | 95 | 95
Not Completed | 3 | 1
Not completed — Adverse Event | 2 | 1
Not completed — Physician Decision | 1 | 0
Period: Period 2: Open-label Period
Arm/Group | Placebo / Teneli + SU | Teneli / Teneli + SU
Started | 95 | 95
Completed | 87 | 85
Not Completed | 8 | 10
Not completed — Adverse Event | 4 | 6
Not completed — Lack of Efficacy | 3 | 1
Not completed — Physician Decision | 0 | 3
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo / Teneli + SU | Teneli / Teneli + SU | Total
Number analyzed (Participants) | 98 | 96 | 194
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (7.8) | 58.4 (8.6) | 59.4 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 34 | 66
  Male | 66 | 62 | 128

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c at Week 12
Description: The change from Baseline in HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at Week 12. Least squares means were derived from an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline HbA1c as a covariate.
Time Frame: at Week 0 and Week 12
Population: The full analysis set, consisting of all type 2 diabetic patients, who received at least one dose of study drug and who had at least one efficacy data after randomization. Analysis based on last observation carried forward, where the last postbaseline double-blind observed value was carried forward and used for Week 12 where data was missing.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo / Teneli + SU | Teneli / Teneli + SU
Number analyzed (Participants) | 98 | 96
percentage of HbA1c | 0.29 (0.06) | -0.71 (0.06)

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 12
Description: The change from Baseline in Fasting Plasma Glucose collected at Week 12. Least squares means were derived from an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline Fasting Plasma Glucose as a covariate.
Time Frame: at Week 0 and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg / dL
Arm/Group | Placebo / Teneli + SU | Teneli / Teneli + SU
Number analyzed (Participants) | 98 | 96
mg / dL | 9.8 (2.2) | -17.3 (2.2)

3. Secondary Outcome: Change From Baseline in the Areas Under the Curve From 0 to 2 h (AUC0-2h) for Postprandial Plasma Glucose at Week 12
Description: The change from Baseline in AUC0-2h for Postprandial Plasma Glucose collected at Week 12. Least squares means were derived from an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline AUC0-2h for Postprandial Plasma Glucose as a covariate.
Time Frame: 0, 0.5, 1, 2 hours post-dose at Week 0 and Week 12
Population: The full analysis set, consisting of all type 2 diabetic patients, who received at least one dose of study drug and who had at least one efficacy data after randomization.
Measure: Least Squares Mean (Standard Error); unit: mg・hr/dL
Arm/Group | Placebo / Teneli + SU | Teneli / Teneli + SU
Number analyzed (Participants) | 92 | 92
mg・hr/dL | 15.514 (6.072) | -65.544 (6.072)

4. Secondary Outcome: Change From Baseline in 2-hour Postprandial Plasma Glucose at Week 12
Description: The change from Baseline in 2-hour Postprandial Plasma Glucose collected at Week 12. Least squares means were derived from an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline 2-hour Postprandial Plasma Glucose as a covariate.
Time Frame: at Week 0 and Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mg / dL
Arm/Group | Placebo / Teneli + SU | Teneli / Teneli + SU
Number analyzed (Participants) | 92 | 93
mg / dL | 6.0 (4.4) | -43.1 (4.4)

ADVERSE EVENTS:
Groups:
- Placebo/Teneli + SU (Data Through Week 12): Placebo for 12 weeks (double-blind period) followed by teneligliptin for an additional 40 weeks (open-label period) in combination with glimepiride. The adverse events which occured from Week 0 to Week 12 were shown.
  MedDRA 13.0
- Teneli/Teneli + SU (Data Through Week 12): Teneligliptin for 12 weeks (double-blind period) followed by teneligliptin for an additional 40 weeks (open-label period) in combination with glimepiride. The adverse events which occured from Week 0 to Week 12 were shown.
  MedDRA 13.0
- Placebo/Teneli + SU (Data From Week 12 to Week 52): Placebo for 12 weeks (double-blind period) followed by teneligliptin for an additional 40 weeks (open-label period) in combination with glimepiride. The adverse events which occured from Week 12 to Week 52 were shown.
  MedDRA 13.1
- Teneli/Teneli + SU (Data Through Week 52): Teneligliptin for 12 weeks (double-blind period) followed by teneligliptin for an additional 40 weeks (open-label period) in combination with glimepiride. The adverse events which occured from Week 12 to Week 52 were shown.
  MedDRA 13.1
Arm/Group | Placebo/Teneli + SU (Data Through Week 12) | Teneli/Teneli + SU (Data Through Week 12) | Placebo/Teneli + SU (Data From Week 12 to Week 52) | Teneli/Teneli + SU (Data Through Week 52)
Serious Adverse Events (participants affected / at risk) | 2/98 | 0/96 | 2/95 | 7/96
Other Adverse Events (participants affected / at risk) | 60/98 | 62/96 | 89/95 | 89/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Teneli + SU (Data Through Week 12) (N=98) | Teneli/Teneli + SU (Data Through Week 12) (N=96) | Placebo/Teneli + SU (Data From Week 12 to Week 52) (N=95) | Teneli/Teneli + SU (Data Through Week 52) (N=96)
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Maculopathy (Eye disorders) | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0
Retinal vein occlusion (Eye disorders) | 0 | 0 | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Loose body in joint (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Ovarian enlargement (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Teneli + SU (Data Through Week 12) (N=98) | Teneli/Teneli + SU (Data Through Week 12) (N=96) | Placebo/Teneli + SU (Data From Week 12 to Week 52) (N=95) | Teneli/Teneli + SU (Data Through Week 52) (N=96)
Body tinea (Infections and infestations) | 0 | 0 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 3 | 8
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 2 | 1
Dermatitis infected (Infections and infestations) | 0 | 1 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 0 | 5 | 2
Gastroenteritis vibrio (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 2 | 1
Impetigo (Infections and infestations) | 0 | 1 | 0 | 1
Infected bites (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 2 | 1 | 2
Nasopharyngitis (Infections and infestations) | 16 | 19 | 26 | 32
Onychomycosis (Infections and infestations) | 0 | 1 | 0 | 2
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 3 | 4 | 11 | 5
Tinea cruris (Infections and infestations) | 0 | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 1 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Infected epidermal cyst (Infections and infestations) | 0 | 0 | 1 | 0
Gingival abscess (Infections and infestations) | 0 | 0 | 0 | 1
Helicobacter infection (Infections and infestations) | 0 | 0 | 1 | 0
Enteritis infectious (Infections and infestations) | 0 | 0 | 1 | 0
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 2 | 12 | 9
Depression (Psychiatric disorders) | 0 | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1
Cervicobrachial syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 2 | 4
Dizziness (Nervous system disorders) | 1 | 0 | 3 | 0
Headache (Nervous system disorders) | 1 | 2 | 1 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 2 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 1 | 0
Carotid arteriosclerosis (Nervous system disorders) | 1 | 0 | 1 | 0
Occipital neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 3 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 3 | 3
Conjunctivitis allergic (Eye disorders) | 2 | 0 | 3 | 0
Diabetic retinopathy (Eye disorders) | 0 | 1 | 3 | 8
Eyelid ptosis (Eye disorders) | 0 | 1 | 0 | 1
Keratitis (Eye disorders) | 0 | 1 | 0 | 1
Trichiasis (Eye disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 1 | 0
Normal tension glaucoma (Eye disorders) | 0 | 1 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 2 | 2
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 2
External ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 2 | 4
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 7 | 9
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2 | 3 | 6
Dental caries (Gastrointestinal disorders) | 1 | 0 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 3 | 4
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 2 | 1
Gastritis atrophic (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gingivitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Periodontal disease (Gastrointestinal disorders) | 2 | 1 | 2 | 4
Periodontitis (Gastrointestinal disorders) | 1 | 1 | 2 | 4
Periproctitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 1 | 3
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 3 | 3
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cutaneous amyloidosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 4 | 6
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Senile pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 3
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hyperkeratosis palmaris and plantaris (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 10
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 3
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 4
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 3
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 2
Feeling abnormal (General disorders) | 0 | 0 | 2 | 0
Malaise (General disorders) | 0 | 0 | 2 | 2
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Thirst (General disorders) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 4 | 3 | 6
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 4
Blood creatine phosphokinase increased (Investigations) | 2 | 2 | 3 | 8
Blood potassium increased (Investigations) | 0 | 2 | 2 | 2
Blood pressure decreased (Investigations) | 0 | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 2 | 3 | 4 | 5
Blood urea increased (Investigations) | 1 | 1 | 0 | 2
Blood uric acid increased (Investigations) | 0 | 2 | 3 | 4
Gamma-glutamyltransferase increased (Investigations) | 0 | 2 | 3 | 3
Glucose urine present (Investigations) | 21 | 2 | 17 | 11
Blood urine present (Investigations) | 3 | 1 | 7 | 6
Platelet count decreased (Investigations) | 0 | 1 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 1 | 1
Protein urine present (Investigations) | 5 | 4 | 13 | 16
Urine ketone body present (Investigations) | 2 | 2 | 2 | 6
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 2
Carotid intima-media thickness increased (Investigations) | 0 | 0 | 0 | 1
Helicobacter test positive (Investigations) | 0 | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 5 | 5
Bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Eye penetration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Nail avulsion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Stab wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 3 | 6
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Open wound (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 3
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ear abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Avulsion fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Loose body in joint (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other